CLINICAL TRIAL: NCT00401388
Title: Sarcoma Alliance for Research Through Collaboration (SARC) Multicenter Trial: A Phase II Trial of Perifosine in Patients With Chemo-Insensitive Sarcomas
Brief Title: A Trial of Perifosine in Patients With Chemo-Insensitive Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Collaborators: Sarcoma Alliance for Research through Collaboration (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 214; NCT00411502 (obsolete NCT alias)
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2012-02

CONDITIONS: Chondrosarcomas; Alveolar Soft Part Sarcomas; Extra Skeletal Myxoid Chondrosarcomas
Keywords: Chemo Insensitive Sarcomas; Chondrosarcomas; Alveolar soft part sarcomas; Extra skeletal myxoid chondrosarcomas; Perifosine
MeSH Terms: conditions — Chondrosarcoma; Sarcoma, Alveolar Soft Part | interventions — perifosine; Loperamide; Allopurinol; Antiemetics

STUDY DESIGN:
Intervention Model Description: One treatment arm: Perifosine. Three groups related to sarcoma subtype: histologically or cytologically confirmed diagnosis of (a) chondrosarcoma, (b) alveolar soft part sarcoma and (c) extra-skeletal myxoid chondrosarcoma.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A: chondrosarcoma (Experimental): Patients with sarcoma subtype: histologically or cytologically confirmed diagnosis of chondrosarcoma.
  Supportive Care Guidelines for perifosine include antiemetic prophylaxis (antiemetics will be administered at the treating investigator's discretion), diarrhea management (loperamide), and hyperuricemia prophylaxis (allopurinol).
  Interventions: Drug: Perifosine; Other: Loperamide; Other: Allopurinol; Other: Antiemetics
- Group B: alveolar soft part sarcoma (Experimental): Patients with sarcoma subtype: histologically or cytologically confirmed diagnosis of alveolar soft part sarcoma.
  Supportive Care Guidelines for perifosine include antiemetic prophylaxis (antiemetics will be administered at the treating investigator's discretion), diarrhea management (loperamide), and hyperuricemia prophylaxis (allopurinol).
  Interventions: Drug: Perifosine; Other: Loperamide; Other: Allopurinol; Other: Antiemetics
- Group C: extra-skeletal myxoid (Experimental): Patients with sarcoma subtype: histologically or cytologically confirmed diagnosis of extra-skeletal myxoid chondrosarcoma.
  Supportive Care Guidelines for perifosine include antiemetic prophylaxis (antiemetics will be administered at the treating investigator's discretion), diarrhea management (loperamide), and hyperuricemia prophylaxis (allopurinol).
  Interventions: Drug: Perifosine; Other: Loperamide; Other: Allopurinol; Other: Antiemetics

INTERVENTIONS:
Drug: Perifosine — Perifosine is available in 50 mg tablets. Patients will take two perifosine 50 mg tablets orally once a day at bedtime with food.
  Other Names: D-21266; KRX-0401
Other: Loperamide — All patients should be instructed to take loperamide at the earliest signs of diarrhea and/or abdominal cramping after beginning perifosine.
Other: Allopurinol — Patients with a known history of hyperuricemia and/or gout should receive prophylactic treatment with allopurinol 300 mg po daily.
Other: Antiemetics — Antiemetic prophylaxis will be administered at the treating investigator's discretion.

SUMMARY:
This is a phase II study of perifosine in patients with chondrosarcomas, alveolar soft part sarcomas and extra-skeletal myxoid chondrosarcomas. Patients will receive perifosine 100 mg orally qhs with food until disease progression. The goals of this study include:

* In this study a daily dose of perifosine previously determined to be relatively non-toxic will be evaluated in patients with chondrosarcomas, alveolar soft part sarcomas and extra-skeletal myxoid chondrosarcomas.
* Response to therapy will be based on regression of measurable disease according to Choi criteria. Time to progression and duration of stable disease will be measured as secondary endpoints of the study.

DETAILED DESCRIPTION:
This is a phase II study of perifosine in patients with chondrosarcomas, alveolar soft part sarcomas and extra-skeletal myxoid chondrosarcomas. Patients will receive perifosine 100 mg orally qhs with food until disease progression.

Perifosine is available in 50 mg tablets. Patients will take two perifosine 50 mg tablets orally once a day at bedtime with food. Administering the drug qhs has been shown to decrease gastrointestinal toxicity in some patients. Patients may need anti-emetics and/or anti-diarrheals. All patients may continue therapy unless disease progression is documented on two occasions at least 4 weeks apart. Patients who experience toxicity may continue on treatment with doses delayed or reduced. Evaluation of all lesions for progression or response will be made at 3-month intervals.

STUDY KEY POINTS

* Treatment will be administered on an outpatient basis in 28-day cycles.
* Growth factors should not be needed, however, use by patients on this trial is NOT prohibited.
* A favorable outcome will be defined as a complete or partial response according to the Choi criteria or stable disease by the Choi criteria for 6 months or longer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of chondrosarcoma, extra-skeletal myxoid chondrosarcoma or alveolar soft part sarcoma.
* Patients may have had prior chemotherapy, but if the patient has had three or more forms of prior chemotherapy for metastases, the patient's clinical course should be discussed with the study chairman before the patient is enrolled on study
* Patients must have progression of disease by Choi criteria.
* ECOG performance status 0-1. Patients with ECOG PS of 2 may be admitted with approval from the study chairman.
* At least 13 years of age.
* Patients must have measurable disease.
* Patients who have brain metastases that have not progressed for at least 2 months following surgery or radiotherapy will be considered after discussion with the study chairman.
* Patients must have a life expectancy of more than 3 months.
* Patients must have normal organ and marrow function, unless in the opinion of the treating investigator, the abnormality is related to tumor, and the study chairman agree the abnormality is unlikely to affect the safety of perifosine use. Normal organ and marrow function is described below:

  * ANC >1.5 x 109 /L
  * Platelets >75,000/ mm3
  * HCT > 28% (with or without growth factor support)
  * Creatinine <= 2.5 mg/dl
  * Total bilirubin < 1.5 x upper limit of normal
  * Transaminase <= 2.5 x upper limit of normal
* Patients must have recovered from acute toxicity related to prior therapy, including surgery or radiotherapy to grade <= 1 (excluding alopecia) at the time of enrollment.
* Patients must be able to ingest oral medications or to obtain them through a gastrostomy tube.
* Female patients who are pregnant or lactating are ineligible. All females of childbearing potential must have a negative urine or serum pregnancy test within 72 hours of treatment. Men and women of childbearing potential must agree to employ adequate contraception to prevent pregnancy while on therapy and for four weeks after the completion of treatment.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients receiving investigational or commercial agents or therapies administered with the intent to treat the patient's malignancy, except bisphosphonates.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine).
* Uncontrolled intercurrent illness-including, but not limited to, ongoing or active infection-and psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment) or New York Heart Assoc. class II-IV congestive heart failure.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-11; Primary Completion 2011-01 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Response rate | >= 6 months
  To investigate whether perifosine has a response rate of > 20% in this group of patients with chemo-insensitive sarcomas.

SECONDARY OUTCOMES:
Best overall response | >= 6 months
  Best response recorded from the start of the treatment until disease progression/recurrence.
Stable disease of six months or greater | >= 6 months
  Stable disease is measured from the start of treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: Dejka Araujo, MD, Study Chair — MD Anderson Cancer Center, Dept of Sarcoma